CLINICAL TRIAL: NCT04299906
Title: Physician-Initiated PMCF Trial Investigating the Solaris Vascular Stent Graft for the Treatment of Iliac Lesions - SOLARIS Peripheral PMCF Trial
Brief Title: SOLARIS Peripheral PMCF Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr. Sabrina Overhagen (Other)
Collaborators: FCRE (Foundation for Cardiovascular Research and Education) (Other); Scitech Produtos Medicos Ltda (Industry)
Responsible Party: Sponsor-Investigator, Dr. Sabrina Overhagen, Study Director, FCRE (Foundation for Cardiovascular Research and Education)
Organization: FCRE (Foundation for Cardiovascular Research and Education) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCRE-191127; NCT04545281 (obsolete NCT alias)
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Peripheral Arterial Disease; Iliac Artery Stenosis; Common Femoral Artery Stenosis
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Solaris Vascular Stent Graft (Experimental): Implant of Solaris Vascular Stent Graft in aorto-iliac lesions
  Interventions: Device: Solaris Vascular Stent Graft

INTERVENTIONS:
Device: Solaris Vascular Stent Graft — Solaris Vascular Stent Graft for treatment of Iliac Lesions

SUMMARY:
The objective of this clinical investigation is to evaluate, in a controlled setting, the long-term (up to 12 months) safety and efficacy of the Solaris Vascular Stent Graft (Scitech) in clinical settings when used according to the indications of the IFU.

ELIGIBILITY:
Inclusion Criteria:

* Corresponding to the IFU indications/contra-indications and according to the current medical guidelines for minimally invasive peripheral interventions.
* Patient presenting with a stenotic or occlusive lesion at the iliac arteries suitable for stenting (on indication for primary stenting, based on the discretion of the investigator)
* Patient presenting a score from 2 to 5 following Rutherford classification
* Patient is willing to comply with specified follow-up evaluations at the specified times for the duration of the study
* Patient is >18 years old
* Patient (or their legal representative) understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* The target lesion is either a modified TASC-II class A, B, C or D lesion.
* The target lesion has angiographic evidence of stenosis or restenosis > 50% or occlusion which can be passed with standard guidewire manipulation
* There is angiographic evidence of a patent Common and Deep Femoral Artery

Exclusion Criteria:

* PTA is technically not possible (not feasible to access the lesion or a defect with the guidewire or balloon catheter)
* Presence of an aneurysm immediately adjacent to the site of stent implantation
* Stenosis distal to the site of stent implantation
* Lesions in or adjacent to essential collaterals(s)
* Lesions in locations subject to external compression
* Heavily calcified lesions resistant to PTA
* Patients with diffuse distal disease resulting in poor stent outflow
* Patients with a history of coagulation disorders
* Patients with aspirin allergy or bleeding complications and patients unable or unwilling to tolerate anticoagulant/antiplatelet therapy and/or non-responders to anticoagulant/antiplatelet therapy
* Fresh thrombus formation
* Patients with known hypersensitivity to the stent material (L605) and/or PTFE
* The target lesion is either a modified TASC-II class B or D lesion with aortic or common femoral lesion involvement.
* Previously implanted stent(s) at the same lesion site
* Reference segment diameter is not suitable for the available stent design
* Untreatable lesion located at the distal outflow arteries
* Use of alternative therapy (e.g. atherectomy, cutting balloon, laser, radiation therapy) as part of the index procedure
* Patients refusing treatment
* Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated
* Patients who exhibit persistent acute intraluminal thrombus of the proposed lesion site
* Perforation at the angioplasty site evidenced by extravasation of contrast medium
* Patients with a history of prior life-threatening contrast medium reaction
* Patients with uncorrected bleeding disorders
* Female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding
* Life expectancy of less than twelve months
* Any planned surgical intervention/procedure within 30 days of the study procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Patient is currently participating in another investigational drug or device study that has not completed the entire follow up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary Patency Rate at 12 month follow-up | 12 months post-op

SECONDARY OUTCOMES:
Primary Patency Rate at 1- and 6 month follow-up | 1 monthand 6 months post-op
Stent Graft Occlusion Rate at pre-discharge, 1-, 6-, and 12-month follow-up | 1day, 1 month, 6 month and 12 month post-op
Ankle-Brachial Index at 1-, 6- and 12-month follow-up compared with baseline ABI | 1-, 6- and 12-month post-op
Amputation rate at 1-, 6- and 12-month follow-up, defined as any amputation above the knee | 1-, 6- and 12-month post-op
Performance success rate at baseline | during procedure
  defined as a composite of (a) successful in sealing acute perforation or rupture; (b) successful in treating aneurysm and fistulae ; (c) restoration of blood flow
in-stent restenosis rate at 1-, 6- and 12-month post-op | 1-, 6-, 12-month post-op
Freedom from Target Lesion Revascularization at 1-, 6- and 12-month post-op | 1-, 6- and 12-month post-op
  defined as freedom from a repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the treated lesion edge
Serious Adverse Events (SAE's) until 12-month post-op | within 12-months post-op
Technical success rate | during procedure
  defined as the ability to achieve final residual angiographic stenosis no greater than 30%
Clinical success at follow-up | 1-, 6- and 12-month post-op
  defined as an improvement of Rutheford Classification at 1-, 6- and 12-month follow-up of one class or more as compared to the pre-procedure Rutherford classification

CONTACTS AND LOCATIONS:
Overall Officials: Michel Bosiers, MD, Principal Investigator — Insel Spital Bern
Locations (10):
- Germany (6):
  - Hospital Hochsauerland, Arnsberg
  - Saarland University Medical Center, Homburg
  - University Hospital Leipzig, Leipzig
  - St. Franziskus Hospital, Münster
  - University Hospital Münster, Münster
  - Hospital Oldenburg, Oldenburg
- Italy (2):
  - Azienda Ospedaliera di Perugia, Perugia
  - Fondazione Policlinico Gemelli, Rome
- Netherlands (2):
  - MCL Leeuwarden, Leeuwarden
  - St. Antonius Hospital, Nieuwegein

IPD SHARING:
Plan to Share IPD: No